CLINICAL TRIAL: NCT06134726
Title: Temporomandibular Joint in Patients With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Syrian Private University (Other)
Responsible Party: Principal Investigator, Diaa Haj Ali, medical doctor Diaa Haj Ali, Syrian Private University
Other Study IDs: BX63413,2021
Record Dates: First submitted 2023-11-03; First posted 2023-11-18 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Temporomandibular Joint Disorders; Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Temporomandibular joints; Bruxism
MeSH Terms: conditions — Temporomandibular Joint Disorders; Arthritis, Rheumatoid; Bruxism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RA group
  Interventions: Diagnostic Test: seropositivity of rheumatoid factor
- Control group
  Interventions: Diagnostic Test: seropositivity of rheumatoid factor

INTERVENTIONS:
Diagnostic Test: seropositivity of rheumatoid factor — All participants were tested for seropositivity of rheumatoid factor and anticitrullinated protein antibodies
  Other Names: anticitrullinated protein antibodies

SUMMARY:
the investigators study aimed to evaluate temporomandibular joint involvement in rheumatoid arthritis patients and healthy individuals 142 participants were recruited in two groups: 72 patients with Rheumatoid Arthritis (RA), and 70 healthy controls. All participants were tested for seropositivity of rheumatoid factor and anticitrullinated protein antibodies. TMD diagnosis was determined according to the standardized and validated diagnostic criteria for TMD (DC/TMD): myalgia, arthralgia, articular disc, displacement, degenerative joint disease, and headache attributed to TMD. Bruxism, a probable sleep and/or awake bruxism diagnosis was determined based on self-report and several clinical findings.

ELIGIBILITY:
* Inclusion criteria included:

  * age > 18 years old
  * individuals who had a minimum of 12 natural teeth.
* Exclusion criteria

  * included: trauma or surgery on the jaw
  * facial nerve paralysis
  * tooth implant
  * scleroderma
  * cerebrovascular accident
  * schizophrenia
  * steroid injection within the last six months.

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 142 participants were recruited in two groups: 72 patients with Rheumatoid Arthritis (RA), and 70 healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Number of patients with prevalence of TMD | 2 years
  patients were interviewed, filled out the questionnaire, and examined
Number of patients with TMD-pain diagnoses | 2 years
  patients were interviewed, filled out the questionnaire, and examined

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Damascus University, Syria, Damascus, Syria

IPD SHARING:
Plan to Share IPD: Undecided